CLINICAL TRIAL: NCT00374439
Title: Promoting Well-being in Teens
Brief Title: Cognitive Behavioral vs. Interpersonal Therapy (IPT) Prevention of Depression in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Judith Garber, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Horowitz Dis
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Depressive Symptoms
Keywords: depression; adolescents; prevention; schools
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Cognitive-behavioral (Experimental): Participants in this arm received a cognitive-behavioral program
  Interventions: Behavioral: Cognitive-behavioral
- Interpersonal Therapy (Experimental): Participants in this arm received a prevention program based on interpersonal therapy for depression
  Interventions: Behavioral: Interpersonal Therapy
- No intervention (No Intervention): Participants in this arm did not receive an intervention, but complete assessments only

INTERVENTIONS:
Behavioral: Cognitive-behavioral — Cognitive-behavioral approach
  Arms: Cognitive-behavioral
Behavioral: Interpersonal Therapy — Interpersonal therapy approach
  Arms: Interpersonal Therapy

SUMMARY:
The purpose of this study is to evaluate the efficacy of a cognitive-behavioral vs. an interpersonal therapy program for preventing depressive symptoms in adolescents.

DETAILED DESCRIPTION:
Hypothesis -- The cognitive-behavioral and interpersonal therapy prevention programs will be significantly better than the no-intervention control group in preventing depressive symptoms measured at post-intervention and at the 6-month follow-up. Gender differences also will be explored.

ELIGIBILITY:
Inclusion Criteria:

* All students in 9th grade Wellness classes who have parental consent

Exclusion Criteria:

* Students without parental consent

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2004-01 (Actual); Primary Completion 2006-01 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Children's Depression Inventory | 9 weeks
  Change in depressive symptoms from baseline to post-intervention at 9 weeks
Center for Epidemiological Studies - Depression scale | 9 weeks
  Change in depressive symptoms from baseline to post-intervention at 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judy Garber, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States